CLINICAL TRIAL: NCT03310151
Title: Does an Imagined Movement Regime Improve Dexterity Following Conservatively Managed Distal Radius Fractures in Older Adults? A Pilot Randomised Controlled Trial
Brief Title: Do Imagined Movements Improve Dexterity in Distal Radius Fractures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Derby (Other)
Collaborators: Aneurin Bevan University Health Board (Other)
Responsible Party: Principal Investigator, Thomas Hughes, Clinical Specialist Physiotherapist (MSc student), University of Derby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRF2017
Record Dates: First submitted 2017-10-06; First posted 2017-10-16 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Radius; Fracture, Lower or Distal End
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with one control and one interventional group
Masking Description: As this is a small, education, non-funded project masking has not been possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Group follows usual care plus imagined movements in a home exercise plan. The exercises will be taught to the subject by reading through an exercise booklet with them, this ensures the advice is standardised. The imagined movement programme will consist of imagined wrist movement in all planes. The frequency of approximately 10-15 minutes, four times a day has been selected as a practical compromise of previous investigations, (Moseley, 2004 and Frenkel et al., 2014), and mirrors routine advice.
  Interventions: Procedure: Imagined movements
- control (No Intervention): Follows usual care

INTERVENTIONS:
Procedure: Imagined movements — Imagined wrist movements, 10-15 minutes, 4 times a day.
  Other Names: Motor imagery
  Arms: Intervention

SUMMARY:
A distal radius fracture is a break at the wrist end of the long bone on the outside of the forearm. It is common, and can cause problems with stiffness, pain and use of the hand and arm for several months. This study is investigating whether imagined movements whilst in the plaster improve dexterity, reduce pain or improve movement when the plaster is removed. As this is a pilot study the aim is to test research and assessment procedure to guide further studies.

Imagined movements involve imagining the wrist moving, without actually moving the wrist. It has been suggested that immobilisation, for example in plaster, can affect the part of the brain responsible for movement and sensation. It has also been suggested that imagined movement can reduce this impact.

This study is investigating subjects over the age of 50 with relatively low impact trauma. Younger subjects and higher velocity injuries will be excluded as this introduces an unwanted variable. Likewise, any fractures requiring surgery, or subjects with pre-existing upper limb injury or deformity will be excluded.

Patients will be invited to participate following their attendance at the local Accident and Emergency department in Newport, South Wales, or the minor injuries department at Ysbyty Ystrad Fawr Hospital, Ystrad Mynach. Sampling will run for approximately 2 months and all participants will be given standard exercises. All participants will attend an appointment at approximately 1 week and be randomised into treatment or control group. The treatment group will be taught imagined movements and be asked to perform these for 10 minutes, four times a day, the control group will continue with standard exercises.

All subjects will attend again for assessment of dexterity, pain and movement after the plaster has been removed, (4-8 weeks dependent on team). This concludes the study.

DETAILED DESCRIPTION:
At initial attendance in Accident and Emergency, subjects that meet the inclusion criteria will be offered an information sheet, and will be asked whether they want to be included in the trial. If they agree, a consent form regarding being contacted about the study and an assessment form will be completed by the advanced nurse practitioner. The forms will be given to the primary researcher and filed securely to comply with The Data Protection Act. All patients, including those who do not wish to participate or don't meet the criteria will be given the standard advice and exercise booklet. This is usual for this group of patients.

The lead researcher will contact each subject within 3 days to discuss the study, and arrange an appointment at 7-10 days to begin the study. This is necessary ethically in order to provide a 'cooling-off' period for the subjects to consider whether they wish to participate. It will also give time for radiology reports to be completed and any subjects with discounted radius fracture can be excluded.

Potential subjects attending the initial appointment at 7-10 days in the outpatient physiotherapy department will be offered the full consent form. Those that do not attend or do not consent will be referred back to Accident and Emergency and return to usual care. Those that consent will be randomised into control or intervention group using a computerised random number generator. The control group will continue with maintenance exercises. Having a control group means that the intervention (imagined movements) can be isolated and tested with greater confidence. This helps to improve the quality of the study and this benefit to the study is believed to outweigh the small risk that having a control group would raise. By having the control group follow usual care as closely as possible further minimises ethical issues and potential risks. All efforts have been made to ensure this but it is recognised that all participants will need to attend two appointments that they would not normally attend on normal care. These are necessary to provide a cooling off period and collect data for the study.

The intervention group will have the same exercises as the control group plus imagined wrist exercises. The exercises will be taught to the subject by reading through the booklet with them, this ensures the advice is standardised. As the intervention is targeting part of the brain involved in the control of movement, high frequency is considered important. The imagined movement programme, is amalgamated from two previous studies and will consist of imagined wrist movement in all planes. The frequency of 15 minutes every waking hour from one study is deemed impractical and another study suggests that 15 minutes of mental practice a day preserved range of motion. Therefore approximately 10-15 minutes, four times a day has been selected as a practical compromise and mirrors routine advice.

An appointment will be arranged as soon as is practically possible, aiming for the same day or day after removal of plaster at approximately 4-8 weeks, (varies between teams). This is to reduce the chance of movement out of plaster affecting the outcome measures.

At the 4-8 week appointment the primary outcome measures of dexterity using the Purdue peg-board, and secondary outcome measures of pain and active wrist range of motion will be measured and recorded in the outpatient physiotherapy department.

The subjects will be randomised into control or intervention group which will reduce selection bias. Only standardised objective outcome measures are being used which reduces the chances of the researcher influencing responses. As this is a small, educational study there is no funding and therefore the researcher will be randomising the participants, providing the exercises, and assessing the outcome measures. It is recognised that this is a potential source of bias as the researcher is not blind to group allocation, however, as this is a pilot study this is felt to be an acceptable weakness and will be recognised in write up. It is also a valuable educational experience for the student researcher to be involved in each part of the study.

Broadly the timetable will be two months of recruitment followed by data collection which will continue for up to eight weeks after recruitment has terminated. Data analysis and interpretation will commence whilst collection is ongoing and continue for approximately two to four weeks. The final reporting and write up will follow this.

Sampling is planned to run for 2 months and all potential subjects meeting the criteria will be given the opportunity to participate. Metrics from the local departments, (after allowing for subjects not consenting or meeting the criteria), suggest this could produce a sample size of around 40. This is difficult to predict but one of the aims of this pilot study is to test these procedures. Recruitment will be initially undertaken by advanced nurse practitioners in Accident and Emergency.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 and over
* Closed distal radius fracture
* Lives within Aneurin Bevan University Health Board geographically

Exclusion Criteria:

* Aged under 50
* Lives outside Aneurin Bevan University Health Board geographically, or unable to attend appointments
* Open distal radius fracture
* Requires surgery to distal radius fracture
* Fracture is subsequently ruled out
* Any additional upper limb injury
* Bilateral wrist fracture
* Unable to give consent
* Unable to follow instructions or speak English
* Pre-existing wrist injury, deformity or neurological impairment of either upper limb
* Subject describes significant emotional and/or psychological trauma at the time of injury

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Dexterity | 4-6 weeks
  Time in seconds using standardised Purdue peg-board

SECONDARY OUTCOMES:
Pain | 4-6 weeks
  Visual analogue scale for pain (x/10)
Active range of motion of the wrist | 4-6 weeks
  Goniometry of wrist (degrees)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Kennedy, Study Director — University of Derby
Locations (1):
- Aneurin Bevan University Health Board, Newport, Gwent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frenkel MO, Herzig DS, Gebhard F, Mayer J, Becker C, Einsiedel T. Mental practice maintains range of motion despite forearm immobilization: a pilot study in healthy persons. J Rehabil Med. 2014 Mar;46(3):225-32. doi: 10.2340/16501977-1263. PMID 24519331
- [Background] Moseley GL. Graded motor imagery is effective for long-standing complex regional pain syndrome: a randomised controlled trial. Pain. 2004 Mar;108(1-2):192-8. doi: 10.1016/j.pain.2004.01.006. PMID 15109523

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT03310151/Prot_SAP_ICF_000.pdf